CLINICAL TRIAL: NCT00482768
Title: Improving Risk Factors for Diabetes Complications in Primary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: R18DK075692 (NIH); R18DK075692 (NIH)
Record Dates: First submitted 2007-06-04; First posted 2007-06-05 (Estimated); Last update posted 2018-03-19 (Actual); Status verified 2011-03

CONDITIONS: Type 2 Diabetes
Keywords: Diabetes, type II; Primary Health Care; Outpatient Care
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Intervention clinics will receive practice facilitation visits at regular intervals over a 12-month period.
  Interventions: Behavioral: Practice Facilitation
- 2 (No Intervention): Control clinics will deliver usual care for patients with diabetes.

INTERVENTIONS:
Behavioral: Practice Facilitation — Clinics in the experimental arm will meet with a trained facilitator to work on change strategies that will improve risk factors for diabetes complications.
  Arms: 1

SUMMARY:
The purpose of this study is to test an intervention in primary care clinics to improve three risk factors for diabetes complications: glucose control, blood pressure and cholesterol. Subjects in the study will be clinic staff and clinicians, not patients. The intervention is Practice Facilitation. Practice facilitation occurs when a trained facilitator meets with a team of staff and clinicians in each practice over a period of several months. Facilitation meetings create time for learning and reflection by members of the team and improves their communication so that they can adopt and implement a strategy to improve patient care

DETAILED DESCRIPTION:
Current control of hemoglobin A1c, blood pressure and lipids among patients with type 2 diabetes in primary care settings is not adequate to prevent complications. Results from an NIDDK funded R34 pilot study conducted by members of this research team suggest that Practice Facilitation is feasible and may improve these risk factors. Practice facilitation occurs when a trained facilitator meets with a team of staff and clinicians in each practice over a period of several months. Facilitation meetings create time for learning and reflection by members of the team and improves their communication so that they can adopt and implement a strategy to improve patient care. The purpose of this study is to use a Practice Facilitation intervention to improve the above three risk factors among patients with type 2 diabetes in small, autonomous primary care practices. This intervention is based on complex adaptive system theory to support the selection, tailoring and implementation of one or more strategies to improve the above 3 risk factors in each intervention practice. Five strategies will be discussed during the facilitation to stimulate change in each practice: a diabetes registry, point-of-care testing of HbA1c and lipids, group clinic visits, improved decision support during the visit, and patient activation prior to each visit. The specific objectives are : 1) To evaluate the effectiveness and sustainability of practice facilitation to improve risk factors for type 2 diabetes complications across a variety of primary care settings; 2) Assess the implementation of the chronic care model(CCM) in response to the intervention; 3) Examine the relationship between communication within the practice team and the implementation of the CCM model; and 4) From the perspective of the organization conducting the intervention and the primary care practice, examine the cost of implementing the intervention relative to risk factor change. The study will be a cluster randomized trial conducted in 40 primary care practices randomized to intervention or control. Data will be collected on all practices and 40 patients in each practice using a multi-method assessment process at baseline, 12 and 24 months. The intervention will be a series of 15 visits to 20 intervention practices by trained facilitators over 12 months. Primary hypotheses will be tested with 12 month outcome data. Sustainability of the intervention will be tested with 24 month data. Insights will be included in a delayed intervention conducted in control practices and evaluated in a pre-post design.

ELIGIBILITY:
Inclusion Criteria:

* Primary care practice with 5 or fewer physicians
* The practice must have seen at least 50 patients with type 2 diabetes in the past 90 days

Exclusion Criteria:

* Practice owned by a large vertically integrated health care system

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2493 (Actual)
Dates: Start 2007-06; Primary Completion 2012-04 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
glycosylated hemoglobin | 36 months

SECONDARY OUTCOMES:
systolic blood pressure | 36 months
LDL-cholesterol | 36 months
Change in risk of coronary heart disease | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Polly H Noel, PhD, Principal Investigator — University of Texas Health Science Center San Antonio
Locations (1):
- University of Texas Health Sciences Center, San Antonio, Texas, United States

REFERENCES:
- [Background] Parchman ML, Pugh JA, Culler SD, Noel PH, Arar NH, Romero RL, Palmer RF. A group randomized trial of a complexity-based organizational intervention to improve risk factors for diabetes complications in primary care settings: study protocol. Implement Sci. 2008 Mar 5;3:15. doi: 10.1186/1748-5908-3-15. PMID 18321386
- [Background] Noel PH, Lanham HJ, Palmer RF, Leykum LK, Parchman ML. The importance of relational coordination and reciprocal learning for chronic illness care within primary care teams. Health Care Manage Rev. 2013 Jan-Mar;38(1):20-8. doi: 10.1097/HMR.0b013e3182497262. PMID 22310483
- [Background] Bowers KW, Robertson M, Parchman ML. How inclusive leadership can help your practice adapt to change. Fam Pract Manag. 2012 Jan-Feb;19(1):8-11. No abstract available. PMID 22335375
- [Background] Culler SD, Parchman ML, Lozano-Romero R, Noel PH, Lanham HJ, Leykum LK, Zeber JE. Cost estimates for operating a primary care practice facilitation program. Ann Fam Med. 2013 May-Jun;11(3):207-11. doi: 10.1370/afm.1496. PMID 23690319
- [Background] Mackey K, Parchman ML, Leykum LK, Lanham HJ, Noel PH, Zeber JE. Impact of the Chronic Care Model on medication adherence when patients perceive cost as a barrier. Prim Care Diabetes. 2012 Jul;6(2):137-42. doi: 10.1016/j.pcd.2011.12.004. Epub 2012 Jan 20. PMID 22264426
- [Background] Arar NH, Noel PH, Leykum L, Zeber JE, Romero R, Parchman ML. Implementing quality improvement in small, autonomous primary care practices: implications for the patient-centred medical home. Qual Prim Care. 2011;19(5):289-300. PMID 22186171
- [Result] Parchman ML, Noel PH, Culler SD, Lanham HJ, Leykum LK, Romero RL, Palmer RF. A randomized trial of practice facilitation to improve the delivery of chronic illness care in primary care: initial and sustained effects. Implement Sci. 2013 Aug 22;8:93. doi: 10.1186/1748-5908-8-93. PMID 23965255
- [Derived] Noel PH, Parchman ML, Palmer RF, Romero RL, Leykum LK, Lanham HJ, Zeber JE, Bowers KW. Alignment of patient and primary care practice member perspectives of chronic illness care: a cross-sectional analysis. BMC Fam Pract. 2014 Mar 29;15:57. doi: 10.1186/1471-2296-15-57. PMID 24678983